CLINICAL TRIAL: NCT03477760
Title: Multi-Drug Resistant Bacteria Carriage After Travel: Comparison Between Patients Who Have Been Hospitalized in a Foreign Country, or Not During the Previous Year
Brief Title: Multi-Drug Resistant Bacteria Carriage After Travel
Status: Completed | Type: Observational
Sponsor: Hopital Lariboisière (Other)
Responsible Party: Principal Investigator, Célia Lloret-Linares, MD PhD, MD, PhD, Hopital Lariboisière
Other Study IDs: MRB after travel
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Beta Lactam Resistant Bacterial Infection (Disorder)

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen stool
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rectal swab for Multi-Drug resistant bacteria — A rectal swab will be performed at admission of patients to look for intestinal carriage of Multi-Drug resistant bacteria

SUMMARY:
During one month, from 1st to 30th November 2016, all patients admitted in one of the medical Dpt of our Hospital (Internal Medicine Dpt, Endocrinology, ICU) will be screened for multi-drug resistant bacteria carriage (after written consent). They will answer to a questionnaire about previous travel in a foreign country during the previous year, hospitalization or not during this travel.

DETAILED DESCRIPTION:
During one month, from 1st to 30th November 2016, all patients admitted in one of the medical Dpt of our Hospital (Internal Medicine Dpt, Endocrinology, ICU) will be screened for multi-drug resistant bacteria carriage (after written consent), regardless a travel in a foreign country during the past year, or not. They will answer to a questionnaire about previous travel in a foreign country during the previous year, hospitalization or not during this travel. The aim of the study will be to compare the rate of carriage of multi-drug resistant bacteria among previous travelers, or not.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in one of the medical Dpt of our Hospital who have travelled in a foreign country during the previous year

Exclusion Criteria:

* patients who were unable to give written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted in one of the medical Dpt of our Hospital who have travelled in a foreign country during the previous year
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Multi-Drug Resistant bacteria carriage rate | At admission in our Hospital
  Multi-Drug Resistant bacteria carriage assessed by rectal swab

CONTACTS AND LOCATIONS:
Overall Officials: Pierre O Sellier, M.D., Ph.D., Study Director — Hopital Lariboisiere
Locations (1):
- URT, Hopital Lariboisiere, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No